CLINICAL TRIAL: NCT06793280
Title: Evaluation of Colonic Perfusion by Indocyanine Green Angiography During Elective Colorectal Surgery: Randomized Controlled Trial
Brief Title: Evaluation of Colonic Perfusion by Indocyanine Green Angiography During Colorectal Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Roma La Sapienza (Other)
Collaborators: Nuovo Ospedale dei Castelli (Unknown); San Giovanni Addolorata Hospital (Other)
Responsible Party: Principal Investigator, Lidia Castagneto Gissey, Professor, University of Roma La Sapienza
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 6608
Record Dates: First submitted 2024-05-06; First posted 2025-01-27 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2025-03

CONDITIONS: Anastomotic Leak
Keywords: anastomotic leak; colorectal surgery; colorectal cancer
MeSH Terms: conditions — Anastomotic Leak; Colorectal Neoplasms

STUDY DESIGN:
Intervention Model Description: An interim analysis incoroporating a futility assessment is designed to assess whether this trial is likely to meet its objective before its completion
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- ICG angiography (Experimental): luorescence angiography is utilized to assess colonic resection margins and colorectal anastomosis, aiming to evaluate colonic blood flow. If the assessment indicates "insufficient" perfusion at the resection margin, the colon is resected once more to ensure satisfactory blood flow.
  luorescence angiography is utilized to assess colonic resection margins and colorectal anastomosis, aiming to evaluate colonic blood flow. If the assessment indicates "insufficient" perfusion at the resection margin, the colon is resected once more to ensure satisfactory blood flow.
  Colonic resection margins and colorectal anastomosis are intraoperatively assessed using fluorescence angiography to evaluate colonic perfusion. If perfusion at resection margin is considered "insufficient" the colon is resected again in order to obtain adequate perfusion.
  Interventions: Procedure: intraoperative ICG angiography
- No ICG angiography (Active Comparator): Subjective visual measures are employed by the surgeon in order to determine anastomotic perfusion.
  Interventions: Procedure: No intraoperative ICG angiography

INTERVENTIONS:
Procedure: intraoperative ICG angiography — Intraoperative ICG angiography to evaluate colonic perfusion
  Arms: ICG angiography
Procedure: No intraoperative ICG angiography — Visual evaluation of colonic perfusion
  Arms: No ICG angiography

SUMMARY:
Despite advancements in technology and improved surgical techniques, the occurrence of anastomotic leakage (AL) after colorectal surgery remains between 4% and 30%. AL is a feared complication associated with significant morbidity and mortality in colorectal surgery, with its causes being multifaceted. Inadequate blood supply to the intestines is believed to be a major contributor to its development. Various methods have been proposed to objectively assess intestinal perfusion beyond the subjective evaluation done by surgeons during surgery. However, these methods face challenges such as poor reproducibility and high costs, limiting their routine use. In recent years, indocyanine green (ICG) angiography has emerged as a tool for assessing organ perfusion in various medical scenarios. However, only one randomized clinical trial has been conducted regarding its use in evaluating colorectal surgery outcomes, which found that while ICG angiography sometimes led to additional bowel resection, it didn't significantly reduce the rate of anastomotic leaks compared to conventional methods. This could be due to the trial's small sample size, potentially reducing its statistical power. This study aims to investigate whether ICG angiography can lower the rate of anastomotic leaks during laparoscopic colorectal cancer surgery, while also examining its impact on resection margins, perioperative morbidity, and mortality rates.

A total of 561 subjects undergoing laparoscopic colorectal surgery for malignancy, will be randomized in 2 arms: A Study Group undergoing ICG angiography (i.e. colonic perfusion is intraoperatively assessed by ICG angiography and level of resection is selected based on the fluorescence) and a Control Group (i.e. resection is performed based on subjective judgment).

ELIGIBILITY:
Inclusion Criteria:

* Age: 18-85 years
* Malignant colorectal tumors
* Elective surgery

Exclusion Criteria:

* Abdomino-perineal resection
* Emergency procedures
* Conversion to open surgery
* No anastomosis
* Multifocal tumors
* Locally advanced cancer (T4)
* Distant metastases (M+)
* Major vasculopathies (previous PE, DVT, abdominal aorta surgery)
* ICG allergy

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 562 (Estimated)
Dates: Start 2023-05-06 (Actual); Primary Completion 2025-05-06 (Estimated); Study Completion 2025-09-06 (Estimated)

PRIMARY OUTCOMES:
Anastomotic leak rate | 90 days

SECONDARY OUTCOMES:
Modification in the level of resection margins (cm) | intraoperative
RCP levels (POD 3, 5) | 5 days
Early complications (30 days) | 30 days
Mortality | 90 days
Hospital re-admissions | 30 days
Operative time | 1 day

CONTACTS AND LOCATIONS:
Locations (1):
- Lidia Castagneto Gissey, Roma, Italy, Italy

IPD SHARING:
Plan to Share IPD: No